CLINICAL TRIAL: NCT06635473
Title: Effect of Intelligent Intervention Strategies on Self-efficacy and Hospital Readiness of Parents of Preterm Infants: a Randomized Controlled Trial
Brief Title: Effect of Intelligent Intervention Strategies on Self-efficacy and Hospital Readiness of Parents of Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Lin Kang, Clinical Professor, Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUMC
Record Dates: First submitted 2024-09-29; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Premature Delivery
MeSH Terms: conditions — Premature Birth | interventions — Coping Skills; Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Routine nursing, discharge education
- intervention group (Experimental): Intelligent interventions to enhance parents' hospital discharge readiness and self-efficacy.
  Interventions: Behavioral: Information support; Behavioral: Stress and coping; Behavioral: Specialist guidance; Other: Social support and interaction; Behavioral: Parentage development

INTERVENTIONS:
Behavioral: Information support — The experimental group was given intervention measures. According to the general data survey, discharge readiness and self-efficacy assessment, parents were divided into low, middle and high discharge readiness groups and low, middle and high self-efficacy groups, respectively, using WeChat mini programs to push different content.
  Arms: intervention group
Behavioral: Stress and coping — According to the results of self-efficacy and anxiety assessment, different interventions were based on different scores. Give encouragement and affirmation to parents with low anxiety and high self-efficacy. Parents with high anxiety and low self-efficacy should push stress relief methods such as mindfulness relaxation therapy in time. And through the wechat mini program to provide parents to respond to the pressure of the problem, the medical staff to give timely feedback.
  Arms: intervention group
Behavioral: Specialist guidance — Carry out offline science popularization education and specialized training, and highly qualified specialist doctors and nurses will train parents, and parents will be assessed after training, and personalized guidance will be given according to the weak points of each parent's assessment.
  Arms: intervention group
Other: Social support and interaction — Support and encouragement for parents continue from admission to discharge, so that parents feel that even after discharge, there are people to accompany and support them.
  Arms: intervention group
Behavioral: Parentage development — Since parents and children are separated during the hospitalization of preterm infants, we will create an environment where parents still play the role of parents, and stimulate parental competence through kangaroo care, parental touch, and breastfeeding.
  Arms: intervention group

SUMMARY:
1. Construct intelligent management intervention plan for parents of preterm infants from hospital to family based on the medical and health system suitable for China's national conditions.
2. Clinical randomized controlled trials were conducted to verify and evaluate the feasibility and application effect of the intervention program.

DETAILED DESCRIPTION:
Based on the previous literature analysis, this study builds an intelligent intervention scheme based on evidence-based methods and theories. Finally, we selected the parents of preterm infants in the neonatology department of a third class hospital in Shantou to carry out a similar experiment to verify the scheme. With data collected at five critical time points and different interventions provided according to baseline data, the study will reveal significant differences in personalized interventions, self-efficacy at different time points, and hospital discharge readiness among parents of preterm infants in the context of intelligent intervention, showing the relationship between self-efficacy and hospital discharge readiness. This study will fill in the single, traditional model of education and provide new perspectives and methods for future research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for premature infants ① gestational age < 37 weeks；② Premature infants admitted to NICU；③ The duration of hospitalization is more than 5 days.
2. Inclusion and exclusion criteria of primary caregivers of preterm infants ① Preterm infants admitted to neonatology and family caregivers of preterm infants with gestational age < 37 weeks. ② Family members who volunteer to undertake primary care tasks. ③ No mental disorders and can carry out normal language communication； ④ ≥18 years old, proficient in WeChat use；⑤ Informed consent has been signed.

Exclusion Criteria:

1. Exclusion criteria for preterm infants ① intrauterine developmental retardation of preterm infants. ② Preterm infants with a history of major surgery. ③ Unplanned discharge, transfer, transfer or death of premature infants.
2. Exclusion criteria for primary caregivers of preterm infants ① There are recent major mental trauma injuries caused by non-hospitalization factors. ② the caregiver suffers from serious diseases of the heart, brain, lung, kidney and other organs. 3. Shedding criteria: Caregivers who voluntarily asked to withdraw for various reasons during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Parental readiness for discharge | Upon admission and 24 hours before discharge
  The Discharge Readiness Scale - Parent Edition This scale was developed by Weiss Equals in 2006 to assess the discharge readiness of parents of hospitalized children aged 0-18 years. The scale consists of 5 dimensions and 29 items. The scale was scored on a Likert 10-level scale, with scores ranging from 0 to 10 for each item (" complete "to" incomplete ") and an overall score ranging from 0 to 290. The higher the score, the higher the parents' readiness to leave the hospital. Cronbach's α coefficient of the total volume table was 0.85, and Cronbach's α coefficient of each dimension (personal status of parents, personal status of children, knowledge, coping ability and expected support) was 0.71, 0.70, 0.85, 0.86 and 0.84, respectively, indicating good reliability. Chinese scholar Chen et al. Sinicized the scale and verified its good reliability and validity.
Parents' self-efficacy | The day of admission, 24 hours before discharge, and 1 month after discharge
  First developed by German clinical and health psychologist Ralf Schwarzer in 1981, the General self-efficacy Scale has been translated into at least 25 languages and is widely used internationally. In this study, the Chinese version of GSEA was adopted, which was jointly revised by Zhang Jianxin and Schwarzer, and has been proved to have good reliability and validity. The scale has one dimension, a total of 10 items, grades 1 to 4, the test subjects according to their actual situation, "completely correct" counts for 4 points, "mostly correct" counts for 3 points, "somewhat correct" counts for 2 points, "completely incorrect" counts for 1 point, all items are positive, the lowest theoretical score is 10 points. The highest score was 40, and the higher the score, the better the general sense of self-efficacy.

SECONDARY OUTCOMES:
Anxiety | The day of admission, 24 hours before discharge, and 1 month after discharge
  Self-rating Anxiety Scales (SAS) The self-rating Anxiety Scales (SAS), compiled by William W.K. Zung in 1971, is a commonly used self-rating tool for adult anxiety symptoms. It includes 20 items and scores are divided into 1 to 4 levels. There are 15 positive items and 5 negative items in the scale. The 15 positive entries were scored as 1, 2, 3 and 4 points in turn, and the 5 reverse entries (5, 9, 13, 17 and 19) were scored as 4, 3, 2 and 1 points. The score of 20 entries is added to obtain the total score, standard score =SAS total score x 1.25 Take the integer part. Less than 50 is classified as no anxiety, 50 to 59 is classified as mild anxiety, 60 to 69 is classified as moderate anxiety, and more than 69 is classified as severe anxiety. Cronbach's α coefficient is 0.931.
Growth and development indicators of premature infants | 1 week, 1 month, 3 months after discharge
  The weight and length of premature infants were measured. Use the same brand weight scale and calibrate it regularly, taking the average of the two measurements as the measurement result.
Readmission rate of preterm infants | One month after discharge
  Whether to be readmitted to hospital.
Parental care ability | The day of admission, 24 hours before discharge, and 1 month after discharge
  Ability to care for premature infants: ability to care for premature infants refers to the ability of parents or primary caregivers to care for premature infants, including care knowledge, care skills, care attitude and other aspects. This study mainly studies the caring ability of parents of preterm infants and adopts the self-assessment questionnaire of family caring ability of preterm infants compiled by Meng Jingwen et al for quantitative measurement. The questionnaire includes 18 items in 3 parts: caring knowledge of preterm infants, caring technology and caring ability, and adopts Likert 5-level scoring method, with no understanding =1 point. Not very clear =2 points, general understanding =3 points, relatively understanding =4 points, very understanding =5 points. The total score is 18 to 90, and the higher the total score, the higher the caring ability. The content validity of the questionnaire was 0.98, and the Cronbach's α value of the questionnaire was 0.958.
Breastfeeding situation | 1 week, 1 month, 3 months after discharge
  Parents were asked about the feeding conditions of preterm infants after discharge, which were divided into three types: (1) exclusive breastfeeding, (2) formula feeding and (3) mixed feeding.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin K, Zhang S, Zhang Z, Zheng W, Chen Z, Lin Z, Zhang H, Lin N. Implementing intelligent nursing interventions to enhance self-efficacy and hospital readiness in parents of preterm infants: a randomised controlled trial protocol. BMJ Open. 2025 Aug 13;15(8):e101498. doi: 10.1136/bmjopen-2025-101498. PMID 40812802